CLINICAL TRIAL: NCT05533840
Title: Establishment and Application of a New Imaging System for Otology Based on Ultra-high Resolution CT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Beijing Tongren Hospital (Other); Beijing Obstetrics and Gynecology Hospital (Other)
Responsible Party: Principal Investigator, Wang, Zhenchang, Vice President, Director of Medical Imaging Center, Beijing Friendship Hospital
Other Study IDs: 2022-1-1111
Record Dates: First submitted 2022-08-30; First posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Hearing Loss; Tinnitus; Vertigo
Keywords: Otology; Medical imaging; Tomography, X-ray; Diagnosis; Resolution
MeSH Terms: conditions — Hearing Loss; Tinnitus; Vertigo; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Age under 18: Participants under the age of 18
  Interventions: Diagnostic Test: ultra-high-resolution computed tomography exams
- Age 18-30: Participants aged 18-30
  Interventions: Diagnostic Test: ultra-high-resolution computed tomography exams
- Age 31-40: Participants aged 31-40
  Interventions: Diagnostic Test: ultra-high-resolution computed tomography exams
- Age 41-50: Participants aged 41-50
  Interventions: Diagnostic Test: ultra-high-resolution computed tomography exams
- Age 51-60: Participants aged 51-60
  Interventions: Diagnostic Test: ultra-high-resolution computed tomography exams
- Age ≥61: Participants aged ≥61
  Interventions: Diagnostic Test: ultra-high-resolution computed tomography exams

INTERVENTIONS:
Diagnostic Test: ultra-high-resolution computed tomography exams — Participants in the age groups undergo ultra-high-resolution computed tomography exam

SUMMARY:
Tinnitus, hearing loss and vertigo are the three major diseases of otology, affecting hundreds of millions of people in our country, and are major health problems. Ear structures and lesions are deeply embedded in the bone, and CT is the preferred examination technique. The key structures of the ear are small and the lesions are hidden. Spiral CT is "not visible" and "undiagnosed" due to insufficient spatial resolution. The ultra-high-resolution CT independently developed by our team has a spatial resolution of 50 μm, which is 6 times higher than that of high-end spiral CT, and solves the problem of "not showing" ear diseases. However, with the transformation of imaging modes and the improvement of display capabilities, the imaging system of helical CT is no longer applicable. It is urgent to carry out systematic research to create matching imaging plans, imaging anatomy standards and disease assessment standards to solve the problem of "undiagnosed". problem. This project plans to build an adult and pediatric imaging solution based on ultra-high-resolution CT to optimize image quality and radiation dose; comprehensively evaluate conduction, sensory, and surgical-related fine structures of the ear, and establish a new 0.1mm-scale image anatomy atlas; A prospective study conducted by the center analyzes the hidden pathological changes of tinnitus, deafness and vertigo, evaluates the diagnostic efficacy of ultra-high-resolution CT for the above diseases, and establishes new diagnostic criteria for lesion detection, symptom correlation, and efficacy evaluation. This project will bring new changes to the practice of otology clinical diagnosis and treatment

ELIGIBILITY:
1. For healthy volunteers

   Inclusion Criteria:
   * Meet the ethical requirements of U-HRCT examination
   * Can cooperate to complete U-HRCT examination
   * There is no relevant medical history in the side ear scanned

   Exclusion Criteria:
   * Clinical symptoms related to middle and inner ear lesions, such as conduction deafness, sensorineural hearing loss, mixed deafness, vertigo, etc.
   * Congenital inner ear malformation
   * Diseases causing bone changes around the middle and inner ear, such as otitis media, tumors , otosclerosis, fibrous dysplasia, etc.
   * history of previous ear surgery and trauma
   * CT image artifacts or incomplete scan coverage
   * incomplete clinical data
2. For patients with otological diseases

Inclusion Criteria:

* Due to tinnitus/deafness/peripheral vertigo/peripheral facial paralysis in the ENT department of our hospital
* Meet the ethical requirements of U-HRCT examination
* Can cooperate with the completion of U-HRCT examination
* Surgery in the ENT department of our hospital
* At least one follow-up or re-examination after discharge

Exclusion Criteria:

* History of previous ear surgery and trauma
* CT image artifacts or incomplete scanning coverage
* Incomplete clinical data

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: * 50 healthy volunteers (100 ears)
  * otological patients 1450 cases (tinnitus>634 ears, hearing loss>634 ears, and vertigo>181 ears)
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Subjective and objective evaluation methods for CT image quality | 2022.1-2024.12
  Image quality (Likert score) and image noise will be combined to report the optimal image quality-noise combination
Radiological anatomy of normal ears based on ultra-high resolution CT | 2022.1-2024.12
  diameters in milimeter
Radiological anatomy of normal ears based on ultra-high resolution CT | 2022.1-2024.12
  angle in degree
Quantitative diagnostic standard for ear diseases based on U-HRCT image | 2022.1-2024.12
  shape and position of conductive and senserineural hearing pathways
Quantitative diagnostic standard for ear diseases based on U-HRCT image | 2022.1-2024.12
  size in milimeter of conductive and senserineural hearing pathways

CONTACTS AND LOCATIONS:
Overall Officials: Zhenchang Wang, Prof., Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
The project team has not decided the ways to share the data.